CLINICAL TRIAL: NCT06280469
Title: Single-operator Versus Double-operator in Single-Balloon Enteroscopy：a Prospective, Multicenter, Non-inferiority, Randomized Controlled Study
Brief Title: Single-operator Versus Double-operator in Single-Balloon Enteroscopy
Acronym: SBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shuhui Liang (Other)
Responsible Party: Sponsor-Investigator, Shuhui Liang, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KY20232298-F-2
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Single-balloon Enteroscopy; Operation
MeSH Terms: interventions — Single-Balloon Enteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilot group (Experimental): endoscope and overtube equipped with a balloon are operated by one endoscopist.
  Interventions: Device: Single-Balloon Enteroscopy
- control group (Experimental): endoscope is operated by one endoscopist and overtube equipped with a balloon is operated by one assistant
  Interventions: Device: Single-Balloon Enteroscopy

INTERVENTIONS:
Device: Single-Balloon Enteroscopy — The inflated balloon is supposed to fix the intestine to the endoscope system.Pushing the endoscope deeper into the small bowel with the balloon and enteroscope.

SUMMARY:
Compared with two-person in single-balloon enteroscopy, one-person single-balloon enteroscopy has the advantages of better observation and treatment of lesions, shorter examination time, saving resources in the endoscopy room, and reducing the postoperative discomfort of the examined person, etc. However, there is no comparative study of one-person and two-person in single-balloon enteroscopy.

DETAILED DESCRIPTION:
The incidence rate of chronic small bowel disease in China is 6.14%. Due to the deep location, large length, tortuous shape and large free degree, the diagnosis and treatment of small bowel disease has always been a major challenge in the clinical work of gastroenterology. Although capsule endoscopy can realize the observation of the whole small intestinal mucosa, it cannot effectively observe in real time the suspicious lesions, much less treatment, and its many difficulties still need to be resolved. Enteroscopy allows for real-time, direct visualization of the small intestine and provide effective treatment, which is an important tool for the diagnosis and treatment of small intestinal diseases. The depth of small bowel insertion and whole small bowel examination rate are important indicators for evaluating enteroscopy. However, due to objective factors, such as lesion location and luminal stenosis, the depth of insertion is a better indicator of the quality of enteroscopy, which is more in line with clinical needs.Currently,the single-balloon enteroscopy, which is now more common in clinical practice, have been designed and optimized for relative ease of operation and a shorter learning curve.Compared with two-person in single-balloon enteroscopy, one-person single-balloon enteroscopy has the advantages of better observation and treatment of lesions, shorter examination time, saving resources in the endoscopy room, and reducing the postoperative discomfort of the examined person, etc. However, there is no comparative study of one-person and two-person in single-balloon enteroscopy.Therefore, we propose to conduct a multicenter, noninferiority, randomized controlled study to explore the effect of single and double operation on single balloon small bowel insertion depth, total small bowel examination rate, and lesion detection rate.

ELIGIBILITY:
Inclusion Criteria:

* age greater than eighteen years;
* Suspected small bowel disease with proposed enteroscopy

Exclusion Criteria:

* patients with a history of small bowel surgery;
* patients who fail to perform bowel preparation as required;
* patients at high risk for esophageal varices with risk of bleeding;
* patients who have not planned a deep small bowel examination before enteroscopy, such as a lesion clearly located in the duodenum, proximal jejunum or terminal ileum;
* patients who are in extremely poor physical condition and are not suitable for general anesthesia, as defined by an ASA score greater than 3;
* Pregnant or lactating women;
* Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum insertion depth | up to 2 years
  The maximum insertion position was recognized as having been reached when the anterior scope could not be advanced further after 30 minutes of repeated attempts without completing full small bowel examination

SECONDARY OUTCOMES:
Total enteroscopy rate | up to 2 years
  Completion of full small bowel examination
Positive findings | up to 2 years
  Finding lesions under endoscopy
Advent events | up to 2 years
  Adverse events include gastrointestinal bleeding, abdominal pain and distension,etc.If an adverse event occurs, it will be handled immediately by the operator.
procedural time | Intraoperative
  Including full operative time, enteroscope insertion time, enteroscope exit time, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Zhao YJ, Dai J, Li XB, Xue HB, Zhang Y, Xiong GS, Ohtsuka K, Gao YJ, Liu Q, Song Y, Fang JY, Ge ZZ. Carbon dioxide insufflation improves the intubation depth and total enteroscopy rate in single-balloon enteroscopy: a randomised, controlled, double-blind trial. Gut. 2014 Oct;63(10):1560-5. doi: 10.1136/gutjnl-2013-306069. Epub 2014 Mar 13. PMID 24626435